CLINICAL TRIAL: NCT07109492
Title: The Role of Mandala Painting Before Surgery on Anxiety and Stress
Brief Title: The Role of Mandala Painting Before Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Niran Çoban (Other)
Responsible Party: Sponsor-Investigator, Niran Çoban, Asst.Prof., University of Yalova
Organization: University of Yalova (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NÇ.AT
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Mandala Painting; Surgery; Nurse's Role

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala painting (Experimental): Pre-surgery (Before Mandala Painting) Pre-surgery (After Mandala Painting - 20 minutes later)
  Interventions: Other: Mandala
- Standard care (No Intervention): Since standard care will be applied to the patients in this group, in order to be parallel with the mandala group, the relevant scale questions will be answered by interviewing the patient 20 minutes before and after going to the operating room.

INTERVENTIONS:
Other: Mandala — Mandala Painting
  Arms: Mandala painting

SUMMARY:
Surgical interventions often cause significant anxiety and stress in patients during the preoperative period. In this study, it is aimed to determine the effect of mandala coloring, a non-pharmacological and art-based intervention, on reducing anxiety and stress levels in individuals scheduled for elective surgery. The universe of the study will consist of patients who will undergo elective surgery between June 2025 and June 2026 in the General Surgery Clinic of Istanbul Sultangazi Training and Research Hospital. Data will be collected using the Introductory Information Form, State Anxiety Inventory (STAI-S), Perceived Stress Scale (PSS), and Physiological Parameters Form (including blood pressure, pulse, respiration rate, and oxygen saturation). One day before surgery, patients who meet the inclusion criteria will be informed about the study and randomized into intervention and control groups using a random number table created with MS Excel software. Patients in the intervention group will perform a 20-minute mandala coloring activity in the preoperative waiting period. Before and after the application, participants' anxiety and stress levels will be evaluated with the STAI-S and PSS, and their physiological parameters will be recorded. Patients in the control group will receive standard preoperative care and will be evaluated at the same time points with the same tools, without any intervention. The study aims to provide evidence for the use of mandala coloring as a simple, low-cost, and effective nursing intervention to reduce preoperative anxiety and stress.

DETAILED DESCRIPTION:
Surgical procedures, although often lifesaving and necessary, are known to trigger significant levels of psychological distress, particularly in the preoperative period. This phase, characterized by uncertainty, fear of anesthesia, and concerns about postoperative outcomes, commonly leads to increased levels of anxiety and stress. Preoperative anxiety is reported in up to 85% of surgical patients and is associated with adverse outcomes such as elevated pain perception, delayed recovery, higher analgesic needs, increased cardiac complications, and lower patient satisfaction. While pharmacological approaches are commonly used, there is growing interest in non-pharmacological and holistic strategies to manage preoperative anxiety and stress effectively.

Among the emerging non-drug interventions, art-based therapeutic activities have gained attention due to their accessibility, affordability, and psychological benefits. One such method is mandala coloring, which involves filling in structured circular designs using colors of the participant's choice. The term "mandala" originates from Sanskrit, meaning "circle," and symbolizes wholeness and balance. According to Carl Jung, mandalas help individuals center themselves and connect with their inner states, offering a calming and integrative experience.

Mandala coloring has been shown to reduce stress and anxiety by directing attention to the present moment, promoting mindfulness, and eliciting meditative-like states. Unlike traditional art therapy, mandala coloring does not require artistic skill and can be easily implemented across various age and educational levels. Studies suggest that coloring mandalas decreases cortisol levels, improves emotional regulation, and enhances psychological well-being in different populations.

Despite its recognized benefits in mental health contexts, limited research exists on the use of mandala coloring specifically in surgical patients during the preoperative period. This study aims to fill this gap by evaluating the effect of a short, structured mandala coloring session on anxiety, stress, and selected physiological parameters among patients awaiting elective surgery.

The study will be conducted between June 2025 and June 2026 at Istanbul Sultangazi Training and Research Hospital's General Surgery Clinic. A total of 60 adult patients who meet the inclusion criteria will be recruited and randomly assigned to either the Mandala Coloring Group (intervention) or the Standard Care Group (control) using a random number table created in MS Excel.

On the day before surgery, participants will be informed about the study and will provide written informed consent. Baseline data will be collected using the Introductory Information Form, the State Anxiety Inventory (STAI-S), the Perceived Stress Scale (PSS), and a Physiological Parameters Form, which includes systolic and diastolic blood pressure, pulse rate, respiratory rate, and oxygen saturation.

Patients in the intervention group will engage in a 20-minute mandala coloring activity using standardized coloring sets in a quiet, preoperative room. Those in the control group will receive routine preoperative care in the same setting, without any additional intervention. Following the intervention period, all participants will undergo the same post-test measurements using the aforementioned tools.

By targeting both psychological and physiological indicators, this study aims to demonstrate that mandala coloring is a practical, low-cost, non-pharmacological approach that can be effectively integrated into routine preoperative nursing care. The findings are expected to contribute to evidence-based surgical nursing practices and support the inclusion of creative, holistic methods in the preparation of patients for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are undergoing elective surgery,
* Cholecystectomy Surgery is planned

  * Age 18 and over,
  * Able to communicate,
  * No wounds or injuries on their hands that would prevent them from painting,
  * Volunteer to participate in the study.

Exclusion Criteria:

* Individuals with a previous psychiatric diagnosis,

  * Those with color blindness or visual perception disorders, Patients over 70 years of age
  * Those taking tranquilizers (anxiolytics, antidepressants, etc.),
  * Those with any health problems that may prevent them from painting (fractures, amputations, etc.),
  * Those who are illiterate,
  * Those with communication disabilities will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Mandala Painting on Anxiety | 12 month
  State Anxiety Inventory: In this study, the "State Anxiety Inventory (STAI-I)" will be used before and after the mandala coloring to assess patients' situational anxiety. The inventory evaluates how individuals feel at a particular moment. It includes 20 items, each scored from 1 (Not at all) to 4 (Completely), reflecting the intensity of the emotion experienced. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 are reverse scored. Total scores range from 20 to 80; higher scores indicate greater anxiety. Additionally, the "Trait Anxiety Inventory (STAI-II)" measures general anxiety independent of specific situations, using a similar 20-item structure with frequency-based responses. The full inventory contains 40 items. High scores on either scale indicate higher anxiety levels. This validated tool enables objective pre- and post-intervention comparison of anxiety states in clinical settings.
The Effect of Mandala Painting on Stress | 12 month
  Perceived Stress Scale (PSS) This scale measures the extent to which a person subjectively perceives certain situations as stressful.The scale is a 5-point Likert format (0 = never; 4 = always) and consists of 4 questions for the positive dimension and 6 questions for the negative dimension. Scores obtained from the scale range from 0 to 40, with scores between 27 and 40 indicating perceived high levels of stress, scores between 14 and 26 indicating perceived moderate levels of stress, and scores between 0 and 13 indicating perceived low levels of stress.
  Translated with DeepL.com (free version) The patient will answer PSS questions before and after the mandala coloring.

CONTACTS AND LOCATIONS:
Overall Officials: NİRAN ÇOBAN, Study Director — University of Yalova
Locations (1):
- Niran Çoban, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mavridou P, Dimitriou V, Manataki A, Arnaoutoglou E, Papadopoulos G. Patient's anxiety and fear of anesthesia: effect of gender, age, education, and previous experience of anesthesia. A survey of 400 patients. J Anesth. 2013 Feb;27(1):104-8. doi: 10.1007/s00540-012-1460-0. Epub 2012 Aug 3. PMID 22864564
- [Background] Mitchell M. General anaesthesia and day-case patient anxiety. J Adv Nurs. 2010 May;66(5):1059-71. doi: 10.1111/j.1365-2648.2010.05266.x. Epub 2010 Mar 9. PMID 20337788
- [Background] Curry, N. A., & Kasser, T. (2005). Can coloring mandalas reduce anxiety? Art Therapy, 22(2), 81-85. https://doi.org/10.1080/07421656.2005.10129441
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Adamatti LC, Bandeira D, Ferreira MB. Risk factors for postoperative anxiety in adults. Anaesthesia. 2001 Aug;56(8):720-8. doi: 10.1046/j.1365-2044.2001.01842.x. PMID 11493233
- [Background] Baran, T., & Demirtaş, A. (2022). Mandala boyama etkinliğinin stresle baş etme ve dikkat düzeyine etkisi. Psikoloji Çalışmaları Dergisi, 42(2), 77-91
- [Background] Spielberger, C. D., Gorsuch, R. L., & Lushene, R. E. (1970). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.